CLINICAL TRIAL: NCT01630681
Title: Uppsala University Psychosocial Care Programme: Internet Based Screening and Stepped Care for Adult Cancer Patients With Anxiety and Depression Symptoms - A Randomized Controlled Trial
Brief Title: Internet Based Screening and Stepped Care for Cancer Patients With Anxiety and Depression Symptoms
Acronym: AdultCan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U-CARE AdultCan
Record Dates: First submitted 2012-05-29; First posted 2012-06-28 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Anxiety; Depression
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based stepped care (Experimental): Internet-based stepped care comprises interactive support (Step 1) and Cognitive Behavioral Therapy (CBT; Step 2). Step 1 starts directly after randomization and extends over a 24 months period. Step 2 extends to a period of ten weeks.
  Interventions: Behavioral: Internet-based stepped care
- Standard care (No Intervention)

INTERVENTIONS:
Behavioral: Internet-based stepped care — Interactive support and Cognitive Behavioral Therapy
  Other Names: Self-help program; Internet-based CBT
  Arms: Internet-based stepped care

SUMMARY:
The aim is to evaluate the effects of Internet based Stepped Care on anxiety, depression and health related quality of life in cancer patients with anxiety and depression symptoms, compared to Standard Care, and to evaluate the health-economic effects of the intervention. The investigators also want to examine the development of anxiety and depression symptoms and health related quality of life in cancer patients without initial symptoms.

The primary hypothesis is that Internet based Stepped Care (I-SC) is more effective in relieving anxiety and depression symptoms in cancer patients, compared to Standard Care (SC). Secondary hypotheses are that less anxiety and depression symptoms also means improved health related quality of life and that I SC is cost-effective or at least cost neutral compared to standard care.

The IT-platform Carebase.se is developed within U-CARE. The platform will be used for delivering of interventions and for collection of all patient reported outcomes. Patients with anxiety or depression symptoms according to the Hospital Anxiety and Depression Scale will be randomized to I SC or SC. Patients with no initial anxiety or depression symptoms will be included in descriptive studies. All patients, in the randomized controlled trial and the descriptive study will followed up during 24 months

I-SC comprises interactive support (Step 1) and Cognitive Behavioral Therapy (CBT; Step 2). Step 1 starts directly after randomization and extends over a 24 months period. Step one comprises web-based patient education including psycho-education and easy interventions strategies employed in CBT. Step 1 also includes a FAQ, a discussion board for patients and a personal diary. Project staff (nurses) is responsible for the FAQ and to moderate the discussion board. The nurses will be supervised by a CBT psychologist. They can also turn to other experts in the project group for advices about how to answer patients' questions.

Patients with remaining anxiety or depression symptoms at 1, 4 or 7 months after randomization will be offered Step 2. Step 2 comprise conventional Internet based CBT for common psychological concerns. The participants' chooses to work with modules that correspond to prioritized concerns, e.g. anxiety or depression. The CBT is structured and manualized and include conventional treatment methods with homework and weekly contacts with the psychologist. Step 2 extends over a 10-week period.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Breast- Colorectal- or Prostate cancer or recurrent Colorectal cancer within 3 months form diagnoses

Exclusion Criteria:

* inability to communicate in Swedish
* Karnovsky performance status < 40
* short expected survival (< 6 month)
* cognitive disability (e.g. dementia or psychosis)
* severe depression or suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in depression | From baseline and 10 months later (after intervention)
  Hospital Anxiety and Depression Scale (HADS) - depression subscale. Range 0-21, >7 is defined as doubtful cases and >10 is defined as clinical cases.
  Montgomery Åsberg Depression Rating Scale (MADRS). Range 0-60 points, >30 is defined as severe depression, >3 at question nr. 9 is defined as suicide risk.
Change in anxiety | From baseline and 10 months later (after intervention)
  Hospital Anxiety and Depression Scale (HADS) - anxiety subscale. Range 0-21, >7 is defined as doubtful cases and >10 is defined as clinical cases.
  Spielberger State-Trait Anxiety Inventory State subscale (STAI-S). Range 20-80.

SECONDARY OUTCOMES:
Change in health related quality of life | From baseline and, 1, 4, 7, 10, 18 and 24 months later (after intervention)
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30), the Breast Cancer module (QLQ-BR23), the Colorectal Cancer module (QLQ-CR29) and the Prostate Cancer module (QLQ-PR25).
Change in Cancer related fatigue (CRF) | From baseline and, 1, 4, 7, 10, 18 and 24 months later (after intervention)
  The Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F)
Change in insomnia | From baseline and, 1, 4, 7, 10, 18 and 24 months later (after intervention)
  Insomnia Severity Index (ISI)
Change in posttraumatic stress | From baseline and, 1, 4, 7, 10, 18 and 24 months later (after intervention)
  Posttraumatic Stress Disorder Checklist - Civilian version (PCL-C)

CONTACTS AND LOCATIONS:
Overall Officials: Louise von Essen, Professor, Study Director — Uppsala University
Locations (3):
- Sweden (3):
  - The hospital i Gävle, Gävle, Gävleborg County
  - Uppsala university hospital, Uppsala, Uppland
  - Västmanlands hospital Västerås, Västerås, Västmanland County

REFERENCES:
- [Derived] Hauffman A, Alfonsson S, Igelstrom H, Johansson B. Experiences of Internet-Based Stepped Care in Individuals With Cancer and Concurrent Symptoms of Anxiety and Depression: Qualitative Exploration Conducted Alongside the U-CARE AdultCan Randomized Controlled Trial. J Med Internet Res. 2020 Mar 30;22(3):e16547. doi: 10.2196/16547. PMID 32224483
- [Derived] Mattsson S, Alfonsson S, Carlsson M, Nygren P, Olsson E, Johansson B. U-CARE: Internet-based stepped care with interactive support and cognitive behavioral therapy for reduction of anxiety and depressive symptoms in cancer--a clinical trial protocol. BMC Cancer. 2013 Sep 11;13:414. doi: 10.1186/1471-2407-13-414. PMID 24024826